CLINICAL TRIAL: NCT04786795
Title: MITE (Compound Azintamide Enteric-coated Tablets) in the Treatment of Dyspepsia After Cholecystectomy: a Multicenter, Randomized, Superior, Parallel Controlled Clinical Study
Brief Title: MITE in the Treatment of Dyspepsia After Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2020-049-2
Record Dates: First submitted 2021-02-24; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-01

CONDITIONS: Patients With Dyspeptic Symptoms After Cholecystectomy
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compound Azintamide Enteric-coated Tablets (Experimental): If dyspeptic symptoms occur after laparoscopic cholecystectomy and are randomized, the experimental group takes Compound Azintamide Enteric-coated Tablets. They were registered before medication and on days 14 and 28 after medication, and gastrointestinal symptoms were assessed at each follow-up visit.
  Interventions: Drug: Compound Azintamide Enteric-coated Tablets
- Oryz-aspergillus Enzyme (Placebo Comparator): If dyspeptic symptoms occur after laparoscopic cholecystectomy and are randomized, the control group takes Oryz-aspergillus Enzyme both Pancreatin Tablet and Ursodeoxycholic Acid Tablets. They were registered before medication and on days 14 and 28 after medication, and gastrointestinal symptoms were assessed at each follow-up visit.
  Interventions: Drug: Oryz-aspergillus Enzyme both Pancreatin Tablet and Ursodeoxycholic Acid Tablets

INTERVENTIONS:
Drug: Compound Azintamide Enteric-coated Tablets — the experimental group takes Compound Azintamide Enteric-coated Tablets.They were registered before medication and on days 14 and 28 after medication, and gastrointestinal symptoms were assessed at each follow-up visit
  Arms: Compound Azintamide Enteric-coated Tablets
Drug: Oryz-aspergillus Enzyme both Pancreatin Tablet and Ursodeoxycholic Acid Tablets — the control group takes Oryz-aspergillus Enzyme both Pancreatin Tablet and Ursodeoxycholic Acid Tablets. They were registered before medication and on days 14 and 28 after medication, and gastrointestinal symptoms were assessed at each follow-up visit
  Arms: Oryz-aspergillus Enzyme

SUMMARY:
To confirm the clinical efficacy of Compound Azintamide Enteric-coated Tablets in the treatment of patients with dyspepsia after cholecystectomy (such as abdominal distension, abdominal pain/abdominal discomfort, diarrhea/fatty stool, early satiety, belching, loss of appetite, etc.) by comparing with positive control drug, to observe its safety, and to evaluate the quality of life of subjects before and after treatment

DETAILED DESCRIPTION:
This study is a multi-center, randomized, superiority and parallel controlled clinical study. Third-party institutions will generate random codes according to random numbers of the software and divide them into two groups (Compound Azintamide Enteric-coated Tablets Group, Oryz-aspergillus Enzyme and Pancreatin Tablet and Ursodeoxycholic Acid Tablets Group) in a ratio of 1:1. Random numbers will be sealed and stored in radiopaque envelopes, which will be managed by a designated person not involved in the specific study.

Specific intervention measures: If dyspeptic symptoms occur after laparoscopic cholecystectomy and are randomized, the experimental group takes Compound Azintamide Enteric-coated Tablets, and the control group takes Oryz-aspergillus Enzyme both Pancreatin Tablet and Ursodeoxycholic Acid Tablets. They were registered before medication and on days 14 and 28 after medication, and gastrointestinal symptoms were assessed at each follow-up visit

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years old, male or female;
2. Patients after laparoscopic cholecystectomy, mainly including cholecystectomy due to cholecystitis, gallstones, gallbladder polyps and other benign gallbladder tumors, non-functioning gallbladder;
3. Dyspeptic symptoms occurred 2 weeks after laparoscopic cholecystectomy, including: abdominal distension, abdominal pain/abdominal discomfort, diarrhea/fatty stool, early satiety, belching, loss of appetite;
4. Signed informed consent, agreed to participate in this study.

Exclusion Criteria:

1. Patients with abnormal liver function and renal function;
2. Patients with severe heart and lung dysfunction;
3. Patients with neurological, mental illness or other reasons can not cooperate with the study;
4. Patients with advanced malignant tumors or other serious wasting diseases, any unstable chronic diseases and acute diseases, interfere with the efficacy evaluation of this study (such as patients undergoing chemotherapy) and the completion of the trial plan;
5. Patients with biliary obstruction, acute hepatitis, etc., do not use the test drugs and control drugs, and allergic to the test drugs and control drugs;
6. Patients who have taken digestive enzymes and cholagogue drugs by themselves;
7. Pregnant and lactating women;
8. Patients who are participating in other clinical trials;
9. Patients who cannot be followed up on time.

Elimination Criteria

1. Failure to take medicine as required, that is,Failure to take medicine or missed doses ≥ 3 times within 1week;
2. Taking other digestive enzymes, cholagogues and prokinetic drugs or drugs affecting digestive enzymes and bile secretion and excretion during the study;
3. Adverse events occur, for the benefit of patients, doctors believe that the drug should not be continued; the results of such cases do not participate in the efficacy statistics, but are related to the safety evaluation.

Drop-out Criteria

1. Cases with adverse events and patients are not willing to continue participating in the study.
2. Cases who voluntarily withdrew consent from the study due to poor efficacy and inconvenience in follow-up.
3. cases lost to follow-up due to various reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Symptom assessment | 28days
  scored according to the severity of symptoms. severity: 0 : asymptomatic.
  1. : The patient can recall symptoms only after being reminded.
  2. : There are symptoms, but it does not affect daily life. 3 points: Symptoms are present, affecting daily life.
Efficacy evaluation | 28days
  symptom score improvement rate = (symptom score before treatment - symptom score after treatment)/symptom score before treatment × 100%.
  Significantly effective: symptom score improvement rate > 75%. Effective: symptom score improvement rate 50% ~ 75% (including 50%). Improvement: symptom score improvement rate of 25% ~ 50% (including 25%). Ineffective: symptom score improvement rate < 25%. Worsening: The symptom score increased after medication. Overall response rate = (number of effective cases + number of significantly effective cases)/total number of cases × 100%.

SECONDARY OUTCOMES:
The incidence of adverse events (AE) | 28days
  Serious adverse events (SAE), such as death or life-threatening, hospitalization or prolonged hospitalization, severe disability or severely impaired organ function, etc. Adverse reaction symptoms are recorded in three levels: mild, moderate and severe, and may be related, may not be related, definitely related, and definitely not related. Mild adverse reactions: The symptoms of adverse reactions are mild and can only be remembered after a doctor's inquiry; severe adverse reactions: the main complaints of adverse reactions are strong, affecting the patient's daily life or the continuation of research; moderate adverse reactions: the severity of adverse reactions is moderate Between degree and severe.
  Adverse reactions include any new complaints of discomfort during the study period. If symptoms only worsen during the study, it is not considered an adverse event. Any adverse events should be actively handled
Quality of life assessment | 28days
  The SF-NDI scale was used to assess the impact of dyspeptic symptoms on the quality of life of subjects before and after treatment
Pharmacoeconomic evaluation | 28days
  Pharmacoeconomics includes cost indicators and pharmacoeconomic evaluation indicators that are ultimately used for analysis. Cost indicators include the total direct costs that patients should bear from the start of enrollment to the 28-day follow-up period. From an individual analysis perspective, they include: 1) laboratory inspection costs; 2) medical care and management costs; 3) disease diagnosis costs; 4) The cost of treatment; 5) The cost of treatment of adverse reactions and complications.
  Pharmacoeconomics evaluation indicators use cost-effectiveness analysis (CEA) to calculate the cost-effectiveness ratio for comparison.